CLINICAL TRIAL: NCT05625685
Title: Accelerating Health Equity Via Just-In-Time Adaptive Interventions (JITAIs): Scalable and High Impact mHealth Precision Smoking Relapse Prevention.
Brief Title: Equitable Smoking Relapse Prevention
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in Principal Investigator Affilation/Role
Sponsor: Bryan W. Heckman (Other)
Collaborators: City of Hope Medical Center (Other); Virginia Tech Carilion School of Medicine and Research Institute (Other)
Responsible Party: Sponsor-Investigator, Bryan W. Heckman, Associate Professor, Meharry Medical College
Organization: Meharry Medical College (Other)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: 1P50MD017347-01 (NIH)
Record Dates: First submitted 2022-11-01; First posted 2022-11-23 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Tobacco Use Disorder; Tobacco Dependence
Keywords: Smoking Cessation; Nicotine Replacement Therapy; Ecological Momentary Assessment; GPS; mHealth; Digital Intervention; Social Determinants of Health
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Will employ two interventions as part of a sequential multiple-assignment randomized trial (SMART).
  First-stage intervention - Participants are randomized to one of two arms, QuitBuddy (a novel smoking cessation app) or Control.
  Participants will be randomized again after reaching a predefined tailoring variable, operationalized as biochemically verified 24h smoking abstinence within 1-week from target quit date (TQD).
  Second-stage intervention - Social determinants of health (SDoH) intervention.
  Participants are randomized to receive either a digital SDoH intervention (powered by findhelp.org and integrated into QuitBuddy) or will receive an emailed list of social service providers in their Zip Code (standard care control).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quitbuddy (Experimental): Participants will be assigned to use a smartphone app (QuitBuddy) that will automatically guide NRT treatment delivery through the integration of ecological momentary assessments (EMA) and GPS into personalized relapse prevention algorithms.
  Interventions: Other: Quitbuddy; Other: SDoH Augmentation; Other: SDoH Control
- Control (Active Comparator): Control is intended to approximate the real-world experience where Participants will use The National Cancer Institute's smartphone app (QuitGuide) and will self-manage NRT treatment delivery based on written instructions.
  Interventions: Other: Control; Other: SDoH Augmentation; Other: SDoH Control

INTERVENTIONS:
Other: Quitbuddy — Participants will be mailed a one week supply of nicotine lozenges as nicotine replacement therapy (NRT) for their upcoming quit attempt, with the ability to order more as needed. Participants will have a set "Target Quit Date" (TQD) set on Day 8 after enrollment, following one week of ad-lib smoking that comprises the pre-TQD EMA/GPS smoking data collection. GPS guided NRT usage prompts, via hotspot algorithms, will be provided to participants in the Quitbuddy Arm. Participants will contribute four weeks of post-TQD EMA/GPS data to capture lapses and NRT use in real-time. Carbon Monoxide (CO) levels will be tested at each of the six post-TQD remote assessments to provide objective verification of smoking status (i.e., 1 day, 1 week, 1 month, 2 month, 3 month, and 6 month abstinence rates). Computerized data collection methods (RedCap) will be used throughout the study to optimize quality assurance.
  Arms: Quitbuddy
Other: Control — Participants will be mailed a one week supply of nicotine lozenges as nicotine replacement therapy (NRT) for their upcoming quit attempt, with the ability to order more as needed. Participants will have a set "Target Quit Date" (TQD) set on Day 8 after enrollment, following one week of ad-lib smoking that comprises the pre-TQD smoking data collection. Participants will contribute four weeks of post-TQD data to capture lapses and NRT use. CO levels will be tested at each of the six post-TQD remote assessments to provide objective verification of smoking status (i.e., 1 day, 1 week, 1 month, 2 month, 3 month, and 6 month abstinence rates). Computerized data collection methods (RedCap) will be used throughout the study to optimize quality assurance.
  Arms: Control
Other: SDoH Augmentation — The SDoH intervention is based on the findhelp.org online platform, with customization to meet the specific needs of the study and communities being served: includes validated SDoH assessments, personalized social needs searching based on priorities, access to the most comprehensive social service database, and a streamlined closed loop referral system that integrates with workflows.
Other: SDoH Control — No SDoH intervention

SUMMARY:
The goal of this clinical trial is to test a GPS (Global Positioning System)-enabled smartphone app (QuitBuddy) in current smokers. The main questions it aims to answer are:

* Is Quitbuddy a good treatment for quitting smoking and "staying quit"?
* Will a second treatment that connects people to help for their social and financial needs improve Quitbuddy?

Participants will:

* get nicotine lozenges in the mail
* check in with the study team to report on their quitting progress after 1 day, 1 week, 1 month, 2 months, 3 months, and 6 months

Researchers will compare Quitbuddy to an app made by the National Cancer Institute to see if Quitbuddy is better for helping people stay quit.

DETAILED DESCRIPTION:
Tobacco smoking is a primary preventable trans-diagnostic risk factor that if targeted more effectively, could reduce a wide range of health disparities in prevalence, severity, treatment efficacy, and mortality across many chronic health conditions (e.g., diabetes, obstructive sleep apnea), reduce treatment complexity/multi-morbidity, and reduce healthcare costs up to 80%. The Southeast, in particular, has an urgent need to disrupt the status quo of tobacco control (<2% The Centers for Disease Control and Prevention (CDC) recommended tobacco control appropriations; highest smoking and mortality) driven in large part through neglected patterns of social determinants of health (SDoH; poverty, access to care) that disproportionately impact racial and ethnic minorities in the form of greater smoking and chronic disease rates, and ultimately nearly a decade of life lost. Unfortunately, only 5% of smoking cessation attempts last at least one year, with lower success among Black smokers even though they smoke at similar rates and intensity, and make more quit attempts. Accordingly, mobile health (mHealth) may have particular utility in addressing racial disparities.

Black smokers show high engagement rates with smartphones to access healthcare and greater adherence to digital interventions, which may facilitate tailoring to meet distinct needs. There is an urgent need to overcome equity gaps, which will require diversity and inclusion of individuals from underrepresented races/ethnicities to identify effective treatments. There is a need for just-in-time adaptive interventions (JITAIs) that 1) can be deployed rapidly (ideally before craving occurs), 2) effectively prevent or attenuate cravings quickly, and 3) are amenable to personalized treatment. Quitbuddy, the automated, yet personalized, JITAI app developed by the investigators, allows patients to prepare for high-risk situations before they arise, effectively promoting abstinence and preventing relapse. The overall goals are to optimize smart algorithms, identify personalized relapse risk, and automatically prompt NRT delivery in a real-time, preemptive manner, upon approaching personalized high-risk locations. Results from a National Institute on Drug abuse (NIDA)-funded (K23) pilot randomized controlled trial demonstrated outstanding usability (top 10% of over 500 apps), acceptability (>80% compliance), and technical feasibility (<10% GPS data loss). The investigators will build upon these promising data by testing effectiveness in a fully powered and rigorous SMART design with diverse representation of underserved populations and meeting community needs for SDoH interventions.

Specific Aims

Aims 1 & 2: Evaluate QuitBuddy and SDoH augmentation intervention effectiveness for smoking cessation and relapse prevention via pragmatic remote SMART design (N=2,090).

Expected Outcome: Superior 6-month biochemically verified abstinence rates for the QuitBuddy and SDoH augmentation interventions, relative to controls.

Exploratory Aims: Test potential moderators/mediators of the effectiveness of the interventions.

This approach integrates for the first time established theories of relapse risk, evidence-based treatment, smartphone/GPS technology, and SDoH. This project offers high-impact solutions to address health disparities across a wide range of chronic diseases that disproportionately affect under-served populations.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years of age
* Smoking at least 10 cigarettes per day for the past year
* Literate in English/Spanish
* Willing to make a NRT-aided quit attempt within the next week

Exclusion Criteria:

* Pregnancy (according to urine pregnancy test)
* Breastfeeding or planning to become pregnant (self-report)
* Recent (past 3 months) cardiovascular trauma: myocardial infarction, stroke (self-report)
* Current use (past 30 days) of alternative tobacco products (e.g., electronic cigarettes, smokeless tobacco) or smoking cessation medications (self-report)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-02 (Estimated); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Abstinence Rate | 24 hours
  Self-report. Participant enters number of cigarettes smoked.
NRT Compliance | 24 hours
  Self report. Participant enters number of nicotine lozenges used.
Cravings | 24 hours
  Self reported number of cravings experienced.
Withdrawal 1-day | Measured one day after a participant's target quit-date.
  Minnesota Nicotine Withdrawal Scale - A nine-item self-report scale for examining the severity of nicotine withdrawal symptoms in a subject. Participants select 0 (none) - 4 (severe) for each of the items. Higher scores correspond to higher perceived severity of withdrawal.
Withdrawal 1-week | Measured one week after a participant's target quit-date.
  Minnesota Nicotine Withdrawal Scale - A nine-item self-report scale for examining the severity of nicotine withdrawal symptoms in a subject. Participants select 0 (none) - 4 (severe) for each of the items. Higher scores correspond to higher perceived severity of withdrawal.
Withdrawal 1-month | Measured one month after a participant's target quit-date.
  Minnesota Nicotine Withdrawal Scale - A nine-item self-report scale for examining the severity of nicotine withdrawal symptoms in a subject. Participants select 0 (none) - 4 (severe) for each of the items. Higher scores correspond to higher perceived severity of withdrawal.
Withdrawal 2-month | Measured two months after a participant's target quit-date.
  Minnesota Nicotine Withdrawal Scale - A nine-item self-report scale for examining the severity of nicotine withdrawal symptoms in a subject. Participants select 0 (none) - 4 (severe) for each of the items. Higher scores correspond to higher perceived severity of withdrawal.
Withdrawal 3-month | Measured three months after a participant's target quit-date.
  Minnesota Nicotine Withdrawal Scale - A nine-item self-report scale for examining the severity of nicotine withdrawal symptoms in a subject. Participants select 0 (none) - 4 (severe) for each of the items. Higher scores correspond to higher perceived severity of withdrawal.
Withdrawal 6-month | Measured six months after a participant's target quit-date.
  Minnesota Nicotine Withdrawal Scale - A nine-item self-report scale for examining the severity of nicotine withdrawal symptoms in a subject. Participants select 0 (none) - 4 (severe) for each of the items. Higher scores correspond to higher perceived severity of withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan W Heckman, Ph.D., Principal Investigator — Meharry Medical College
Locations (1):
- Meharry Medical College, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No